CLINICAL TRIAL: NCT03769012
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Ability of Beta-glucan (to Augment Immune Function, Decrease URTI Incidence Rates, and Counter Immune Changes in Marathon Runners
Brief Title: Ability of Beta-glucan Supplementation to Augment Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19BIHK
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2018-12

CONDITIONS: Cold; Cold Symptom; Flu; Flu Symptom; Supplement; Stress; Gastrointestinal Tolerance
MeSH Terms: conditions — Common Cold; Influenza, Human | interventions — beta-Glucans

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, placebo-controlled, parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization schedule will be created and provided to the Investigator indicating the order of randomization. Each participant will be assigned a randomization code according to the order of the randomization list generated using www.randomization.com. Enrolled participants will be randomized to the different treatment arms at day -14. Concealment of the allocation of treatment will be employed through the use of opaque sealed envelopes, each labeled with a randomization number. Each envelope will contain information regarding the treatment associated with each randomization number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Beta-Glucan
  Interventions: Dietary Supplement: Beta-Glucan
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-Glucan — 95% beta-glucan sourced from whole cell Euglena Gracilis
  Arms: Treatment
Dietary Supplement: Placebo — microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This proposed study is designed to assess the efficacy of a capsule containing beta-glucan taken orally daily as compared to a placebo capsule on the URTI symptoms, and the immune response change in marathon runners

DETAILED DESCRIPTION:
At screening, an informed consent form will be given to the potential volunteer. They will be required to read the information and will be given the opportunity to seek more information if needed or provided with the option of taking the consent form home to review prior to making their decision. If agreeable, the volunteer will sign the consent form and receive a duplicate of the signed copy. Once consent has been obtained, the screening visit will proceed. Each volunteer will be sequentially assigned a screening number to be entered in the screening and enrollment log. Screening assessments include: review medical history, assess inclusion and exclusion criteria, vitals, study diary, URTI symptom questionnaire, bowel diary, and GI symptom questionnaire.

The next visit will be scheduled 14 days prior to their marathon date (baseline). Participants will be reminded to complete URTI questionnaire, daily study diary, modified GI symptoms and bowel diary in advance of this baseline visit. At baseline participants will begin daily completion of study diaries, URTI questionnaires, daily bowel diaries, and GI tolerance questionnaires. In clinic subjects will complete mood and stress questionnaires, and blood sample for the analysis of CRP and NK cell activity. In addition, on the day of the marathon the participant will be instructed to complete a muscle soreness assessment.

Two and four weeks post-marathon participants will return to the clinic for with unused investigational product, completed study diaries, daily URTI questionnaires, daily bowel diaries, and GI tolerance questionnaires. In clinic subjects will complete mood and stress questionnaires, and blood sample for the analysis of CRP and NK cell activity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females 21-65 years age
2. Body Mass Index (BMI) > 18 kg/m2 to < 34.99 kg/m2
3. Willing to wash-out for nutritional supplements known to affect immune function
4. Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
5. Agree to keep lifestyle habits consistent
6. Currently registered to participate in a full marathon and on a training regimen
7. Healthy as determined by laboratory results, medical history, and physical exam
8. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the occurrence of the trial
2. Verbal confirmation of previous major gastrointestinal surgery or other major digestive disorder which may interfere with the absorption of nutrients
3. Participant has a known allergy to the test material's active or inactive ingredients
4. Chronic consumption of beta-glucan supplements
5. Consumption of anti-inflammatory medications known to affect immune function
6. On antibiotics within 4 weeks of baseline
7. Currently taking antipsychotic medications
8. Prebiotics and probiotics unless on a stable regimen
9. Verbal confirmation of Type I or Type II diabetes or clinically important renal, hepatic, cardiac, pulmonary, pancreatic, neurologic, or biliary disorder, or cancer to be assessed by QI
10. Verbal confirmation of a diagnosed chronic inflammatory condition
11. Verbal confirmation of autoimmune disease or if immune-compromised
12. Chronic recurring respiratory signs and symptoms due to allergies (including seasonal allergies) or chronic bronchitis, asthma, or wheezing
13. Current or history (within past 6 months) of tobacco use
14. Consumption of >14 standard alcoholic drinks per week

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Global Cold/Flu Symptom Severity Score Wisconsin Upper Respiratory Symptom Survey (WURSS) | ANOVA with 2 and 4 weeks post-marathon
  AUC for cold/flu symptoms from Wisconsin Upper Respiratory Symptom Score

SECONDARY OUTCOMES:
URTI Cold/Flu Symptoms from Wisconsin Upper Respiratory Symptom Survey | ANOVA with 2 and 4 weeks post-marathon
  Total number of symptoms
Severity of cold/flu symptoms from Wisconsin Upper Respiratory Symptom Survey | ANOVA with 2 and 4 weeks post-marathon
  Total severity score (each symptom scored on scale of 0-no symptom to 7-severe symptom)
URTI Episodes from Wisconsin Upper Respiratory Symptom Survey | ANOVA with 2 and 4 weeks post-marathon
  Total number of URTI Episodes/person
Sick days | ANOVA with 2 and 4 weeks post-marathon
  Total number of sick days/person
Sick days | ANOVA with 2 and 4 weeks post-marathon
  Percentage of subjects with sick days
Stress Level from the perceived stress scale | ANOVA with 2 and 4 weeks post-marathon
  Change from baseline on the Perceived Stress Scale
C-Reactive Protein | ANOVA with 2 and 4 weeks post-marathon
  Change in concentration from baseline
Natural Killer Cell Activity | ANOVA with 2 and 4 weeks post-marathon
  Change from baseline
Gastrointestinal symptoms | ANOVA with 2 and 4 weeks post-marathon
  Total gastrointestinal symptom rating score (GSRS)

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No